CLINICAL TRIAL: NCT02637947
Title: A Prospective, Multi-center, Post Market Randomized Controlled Trial Comparing VT Ablation Outcomes Using Remote MAGNETIC Navigation Guided Substrate Mapping and Ablation Versus Manual Approach in a Low LVEF Population
Brief Title: Comparison of VT Ablation Outcomes Using Remote MAGNETIC Navigation Versus Manual Approach in a Low LVEF Population
Acronym: MAGNETIC-VT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In the post-market environment, the RCT design did not allow achievement of enrollment goals
Sponsor: Stereotaxis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-021
Record Dates: First submitted 2015-12-04; First posted 2015-12-22 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Tachycardia, Ventricular
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnetic navigation (Experimental): Catheter ablation using magnetic navigation for ventricular tachycardia via remote magnetic navigation of a NaviStar RMT ThermoCool catheter, or other magnetically compatible catheter, via Stereotaxis's Niobe ES system.
  Interventions: Device: catheter ablation using magnetic navigation
- Manual navigation (Active Comparator): Catheter ablation using manual navigation for ventricular tachycardia via a manually navigated Thermocool catheter, or equivalent catheter.
  Interventions: Device: catheter ablation using manual navigation

INTERVENTIONS:
Device: catheter ablation using magnetic navigation — elimination of cardiac arrhythmias through heating and destroying heart tissue with faulty electrical pathways through the use of Stereotaxis's Niobe ES System with the NaviStar RMT ThermoCool catheter or other magnetically compatible catheters.
  Arms: Magnetic navigation
Device: catheter ablation using manual navigation — elimination of cardiac arrhythmias through heating and destroying heart tissue with faulty electrical pathways through the use of the NaviStar ThermoCool catheter or other manually navigated catheters.
  Arms: Manual navigation

SUMMARY:
The study purpose is to demonstrate that ventricular tachycardia (VT) ablation using the Niobe™ ES system results in superior outcomes compared to a manual approach in subjects with ischemic scar VT in a low ejection fraction population.

DETAILED DESCRIPTION:
This study is a randomized, single-blind, prospective, multi-center post market evaluation. Subjects will be screened for study eligibility and asked to complete written informed consent prior to any study specific testing assessments. After completing written informed consent, a total of 386 subjects will be randomized on a 1:1 basis to receive VT ablation treatment using either the Niobe ES or standard manual catheter ablation treatment using commercially available products. This will be the largest randomized VT study comparing outcomes from RMN to manually guided catheter ablation procedures. Subjects will be randomized according to a computer-generated randomization scheme. Randomization will be blocked at the study site level and subjects will be blinded to group assignment. Since quality of life measurements will be collected during follow-up, this study is single-blinded in order to mitigate patient bias. Clinical evaluations will not be masked to the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* subject has had an ICD previously implanted
* subject has drug-refractory monomorphic VT
* subject is a candidate for ischemic VT RF ablation
* subject has had a myocardial infarction
* subject has a LVEF less than or equal to 35%

Exclusion Criteria:

* subject has non-ischemic VT
* subject has a history of stroke within 1 month prior to enrollment
* subject has had an acute myocardial infarction within 30 days prior to enrollment
* subject has unstable angina
* subject has undergone cardiac surgery within 60 days prior to enrollment
* subject is pregnant or nursing
* subject has a limited life expectancy of 1 year or less (Subjects requiring LVAD/IABP intraprocedural support may be enrolled as long as life expectancy is at least 1 year following the ablation procedure.)
* subject is unable or unwilling to cooperate with study procedures
* subject has a known presence of intracardiac thrombi as determined by echocardiography
* subject has a major contraindication to anticoagulation therapy or coagulation disorder
* subject has had a previous pericarditis or cardiac tumor
* subject has had previous thoracic radiation therapy
* any other reason the investigator considers the subject ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-01; Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
freedom from any VT in the overall cohort | 12 months

SECONDARY OUTCOMES:
acute success of procedure | at end of procedure (immediate)
  non-inducibility of clinical VT and/or other monomorphic VT using typical stimulation protocol for induction
freedom from VT in large scar subpopulation | 12 months
major adverse events | 48 hours post-procedure
  death, cardiac tamponade, stroke, bleeding requiring surgical intervention, progressive heart failure related to VT/VF recurrence
mortality rate | 12 months

OTHER OUTCOMES:
Total number of appropriate ICD defibrillator shocks | 12 months
Total number of ICD applications of anti-tachycardia pacing | 12 months
Total procedure time (skin to skin) | through end of acute procedure, an average of 3 hours
Total fluoroscopy time | through end of acute procedure, an average of 3 hours
Total fluoroscopy dose | through end of acute procedure, an average of 3 hours
Total mapping time | through end of acute procedure, an average of 3 hours
Total ablation time | through end of acute procedure, an average of 3 hours
Total mapping points prior to ablation | through end of acute procedure, an average of 3 hours
Total ablation energy delivery | through end of acute procedure, an average of 3 hours
  Watts X seconds / Total scar surface area
Patient quality of life (SF-12) | 12 months
  Medical Outcomes Study 12-item Short-Form Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (16):
- United States (8):
  - Florida Hospital, Orlando, Florida
  - Augusta University, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Weill Cornell Medical, New York, New York
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Intermountain Heart Institute, Murray, Utah
- Westmead Hospital, Westmead, New South Wales, Australia
- Belgium (2):
  - AZ Sint-Jan, Bruges, West Flanders
  - ZNA Middelheim, Antwerp
- Na Homolce Hospital, Prague, Czechia
- Rigshospitalet, Copenhagen, Denmark
- Chu De Nancy - Hôpitaux De Brabois, Nancy, France
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Derived] Di Biase L, Tung R, Szili-Torok T, Burkhardt JD, Weiss P, Tavernier R, Berman AE, Wissner E, Spear W, Chen X, Neuzil P, Skoda J, Lakkireddy D, Schwagten B, Lock K, Natale A; MAGNETIC VT investigators. MAGNETIC VT study: a prospective, multicenter, post-market randomized controlled trial comparing VT ablation outcomes using remote magnetic navigation-guided substrate mapping and ablation versus manual approach in a low LVEF population. J Interv Card Electrophysiol. 2017 Apr;48(3):237-245. doi: 10.1007/s10840-016-0217-3. Epub 2017 Jan 7. PMID 28064433